CLINICAL TRIAL: NCT00584272
Title: Retrospective Study on the Outcome of Cleft Palate Repair: Comparing US Surgical and Ethicon Suture Materials
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 200715210
Record Dates: First submitted 2007-12-26; First posted 2008-01-02 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Cleft Palate
Keywords: cleft palate; suture materials
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Investigator initiated retrospective chart review to study the effects of changing suture material on the healing and outcome of cleft palate surgery were.

DETAILED DESCRIPTION:
This study aims to show what the effects of changing suture material were on the healing and outcome of cleft palate surgery. The study will be considered successful if we find that either there is an effect on the healing after surgery, one of the suture materials seems to promote better healing and final outcome, or that there is no difference between the suture materials.

ELIGIBILITY:
Inclusion Criteria:

* Cleft palate repair performed at UCDMC between 1/1996 and 6/2006

Exclusion Criteria:

* Those who do not meet the inclusion criteria

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: UCDMC pediatric clinic
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2007-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig W. Senders, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States